CLINICAL TRIAL: NCT03441841
Title: A Cross-over Study of Pharmacokinetic Interaction Comparing Nanoencapsulated Gel of Prilocaine (2.5%), Lidocaine (2.5%) and Association of Prilocaine + Lidocaine 2.5% (Nanorap®) Topically in Healthy Volunteers.
Brief Title: Pharmacokinetic Study of Nanoencapsulated Gel of Lidocaine, Prilocaine and Combination of Lidocaine and Prilocaine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Collaborators: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Principal Investigator, Gilberto De Nucci, Doctor, Galeno Desenvolvimento de Pesquisas Clínicas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GDN 002/16
Record Dates: First submitted 2018-02-10; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Topical Anesthesia
Keywords: local anesthetics; pharmacokinetics; nanotechnology
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine; Prilocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine + prilocaine (Experimental): Single topical dose of a combination of nanoencapsulated lidocaine (2.5%) and prilocaine (2.5%) formulation in a delimited area of 16 cm2 in the volar surface of the forearm.
  Interventions: Drug: Lidocaine + Prilocaine
- Lidocaine (Active Comparator): Single topical dose of lidocaine nanoencapsulated gel (2.5 %) formulation in a delimited area of 16 cm2 in the volar surface of the forearm.
  Interventions: Drug: Lidocaine
- Prilocaine (Active Comparator): Single topical dose of prilocaine (2.5 %) nanoencapsulated gel formulation in a delimited area of 16 cm2 in the volar surface of the forearm.
  Interventions: Drug: Prilocaine

INTERVENTIONS:
Drug: Lidocaine + Prilocaine — Single topical dose of 2g lidocaine + prilocaine 2.5 % formulation.
  Other Names: Nanorap®
  Arms: Lidocaine + prilocaine
Drug: Lidocaine — Single topical dose of 2g lidocaine 2.5 % formulation.
  Arms: Lidocaine
Drug: Prilocaine — Single topical dose of 2g prilocaine 2.5 % formulation.
  Arms: Prilocaine

SUMMARY:
This trial evaluated the pharmacokinetic interaction between fixed doses of lidocaine (2.5%), prilocaine (2.5%) or the association of both (Nanorap®) in healthy volunteers. The drug safety and tolerability was also evaluated.

DETAILED DESCRIPTION:
This study was performed as a monocentric, open, randomized, double-blind, with 3 treatment regimen (lidocaine, prilocaine, or Nanorap®) in 3 periods design. Volunteers were submitted to clinical and laboratory examination before enrollment. Treatments were carried out on 3 different days with a washout period of 7 days between each dose.

After a fasting period (8 h), volunteers received topically 2g of the formulation in a delimited area of 16 cm2 in the volar surface of the forearm. The product was applied to the left arm and venous blood was collected from the right arm. The remaining product was removed with a cotton swab 10 minutes after application. Blood samples (3.5 mL) were collected into heparinized tubes before (0:00) and at 1.0, 2.0, 3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, 9.5, 10.0, 10.5, 11.0, 12.0, 14.0, 16.0 and 24.0 h after the hydrogel application.

Blood samples were centrifuged at 2000 g (4 ⁰C) for 10 minutes and the obtained plasma samples were stored at -20 °C until analysis.

Following dosing, volunteers were monitored for 36 h in a clinical setting safety and tolerability (signs, symptoms, adverse events, and laboratory parameters). The vital signs (blood pressure and pulse rate) were evaluated. ECGs were obtained before (30 min) and at drug Cmax (6 h) for each product application. QT interval corrected by heart rate (QTc) data were obtained from a Bionet Cardiocare 2000 and BMS-Plus software program, using Bazett's formula: QTc = QT/(sqrt RR Interval).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers over 18 years old
* Body mass index (BMI) ≥ 19.0 kg/m² and ≤ 28.75 kg/m²
* No evidence of significant diseases, that, at the investigator's discretion, may affect the participation in the clinical trial, in accordance with the protocol requirements
* Ability to understand the nature and the objective of the clinical trial,including the risks and possible side effects; intention to cooperate with the investigator and act in accordance with the protocol requirements, as confirmed by the informed consent form signature.

Exclusion Criteria:

* Subjects with known hypersensitivity to the compounds of the investigational products, severe allergies or multiple drug allergies
* Existing diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the drug
* Screening laboratory tests presenting deviations deemed as clinically significant, which, due to possible risks, prevents the participation in clinical trial.
* Use of maintenance therapy with any drug
* Drug or alcohol dependence
* Volunteers who ingests more than 5 cups of coffee or tea per day and/or smoke
* Volunteers with unusual eating habits, e.g, vegetarian
* Treatment, within 3 months prior to the initiation of the clinical trial treatment, with any drug known to have a well-established toxic potential to major organs.
* Use of regular medication within 2 weeks before the start of treatment and the date of evaluation, or made use of any medication within one week, except for oral contraceptives or cases where, based on the half-life of the drug and/or active metabolites, complete elimination can be assumed
* Treatment within 6 months prior to the study with any known drug of have a well-defined toxic potential in large organs
* Hospitalization for any reason up to 8 weeks before the start of the treatment of this study
* Participation in a clinical trial during the last 6 months
* Blood donation or other blood loss of more than 450 mL within the last 3 months
* Pregnant, delivery or abortion in the 12 weeks prior to the planned hospitalization
* The volunteer who has any condition that prevents him from participating in the study by judgment of the investigator

Ages: 19 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-02-28 (Actual); Primary Completion 2016-03-19 (Actual); Study Completion 2016-05-06 (Actual)

PRIMARY OUTCOMES:
Measurement of lidocaine and prilocaine plasma levels | 0-24 h
  Blood sampling for the determination of plasma levels of lidocaine and prilocaine in participants of each treatment group.
Maximum Plasma Concentration (Cmax) of lidocaine and prilocaine | 0-24 h
  Determination of Cmax for lidocaine and prilocaine based on plasma concentrations of samples obtained.
Area Under the Curve (AUC) of lidocaine and prilocaine | 0-24 h
  Determination of AUC for lidocaine and prilocaine based on plasma concentrations of samples obtained.

SECONDARY OUTCOMES:
Number of adverse events per participant | Up to 36 h after treatment
  Determination of the number of adverse events, in each treatment group, including clinically relevant alterations of vital signs and laboratory tests results.

CONTACTS AND LOCATIONS:
Locations (1):
- Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No